CLINICAL TRIAL: NCT02527538
Title: Pleth Variability Index Predicts Hypotension in Beach Chair Position in Mechanically Ventilated Adults During General Anesthesia
Brief Title: Prediction of Hypotension During Beach Chair Position Using Pleth Variability Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Chongwha Baek, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Other Study IDs: C2013209(1169)
Record Dates: First submitted 2015-07-28; First posted 2015-08-19 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-08

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pleth: The masimo probe is attached on the index fingertip and cover with black cover in all patients. Record the pleth variability index and blood pressure
  Interventions: Device: Pleth

INTERVENTIONS:
Device: Pleth — apply the masimo probe on index fingertip and record the pleth variability and blood pressure during beach chair position
  Other Names: Masimo

SUMMARY:
The beach chair position for shoulder operation induces hypotension during general anesthesia. Hypotension is induced by decreased preload and contractility due to anesthesia. Masimo is a pulse oximetry which shows pleth variability index noninvasively. The pleth variability may predict the hypotension during beach chair position.

DETAILED DESCRIPTION:
The beach chair position for shoulder operation induces hypotension during general anesthesia. Hypotension is induced by decreased preload and contractility due to anesthesia. Masimo is a pulse oximetry which shows pleth variability index noninvasively. The investigators put the masimo probe before general anesthesia and recorded the values before and after beach chair position, The values include arterial pressure, heart rate, blood pressure, perfusion index, pleth variability index.

The primary end point was the predictive value and threshold or pleth variability index for hypotension induced by the beach chair position. The occurrence of hypotension was counted by using vasopressor. The use of vasopressor was performed when mean blood pressure less than 65 mmHg or 20% of baseline.

The investigators planned to recruit 57 patients.

ELIGIBILITY:
Inclusion Criteria:

* elective shoulder surgery under general anesthesia

Exclusion Criteria:

* right heart failure
* morbid obesity (BMI > 30)
* arrhythmia on preoperative electrocardiography
* pulmonary hypertension
* peripheral vascular disease or pulmonary disease
* pregnant

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age between 20 and 70 years who is planning to undergoing elective shoulder surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
occurrence of hypotension defined as mean blood pressure less than 65 mmHg or 20% of baseline | 10 minutes after beach chair position
  hypotension occurs or not after beach chair position and hypotension was defined as mean blood pressure less than 65 mmHg or 20% of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chongwha Baek, Ph.D., Study Director — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine : Chung-Aung University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siswojo AS, Wong DM, Phan TD, Kluger R. Pleth variability index predicts fluid responsiveness in mechanically ventilated adults during general anesthesia for noncardiac surgery. J Cardiothorac Vasc Anesth. 2014 Dec;28(6):1505-9. doi: 10.1053/j.jvca.2014.04.010. Epub 2014 Aug 29. PMID 25169895